CLINICAL TRIAL: NCT07037524
Title: Prospective Pilot Single-center Study to Evaluate the Safety and Efficacy of Low-dose Radiotherapy in Patients With Heart Failure
Brief Title: Low Dose Radiotherapy for Heart Failure
Acronym: RadioCardio
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Hospital do Coracao (Other)
Collaborators: Financiadora de Estudos e Projetos (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RadioCardio
Record Dates: First submitted 2025-06-17; First posted 2025-06-25 (Actual); Last update posted 2025-06-25 (Actual); Status verified 2025-06

CONDITIONS: Heart Failure - NYHA II - IV
Keywords: Heart Failure; Radiotherapy
MeSH Terms: conditions — Heart Failure | interventions — Radiotherapy

STUDY DESIGN:
Intervention Model Description: Prospective single-center
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single arm (Experimental): Low Dose Radiotherapy
  Interventions: Radiation: Radiation Therapy

INTERVENTIONS:
Radiation: Radiation Therapy — Low single-dose wholw-heart radiotherapy

SUMMARY:
The primary goals of this clinical trial are to evaluate the safety and efficacy of a low dose whole-heart radiotherapy with a single fraction in ten participants with advanced heart failure.

DETAILED DESCRIPTION:
The primary objectives of this prospective phase I/II, single-center study, are to evaluate the safety and efficacy of low dose whole-heart radioherapy (RT) in ten patients with heart failure (HF).

Eligible patients must have clinical-laboratory diagnosis of New York Heart Association grade II or III chronic systolic HF with ejection fraction < 40% and refractoriness to standard clinical treatment defined as the persistence of signs and symptoms of HF despite optimized drug therapy.

All subjects will receive whole-heart RT for a single-dose of 5 Gy. The primary efficacy endpoint will be determined by evaluating the impact of RT on left ventricular ejection fraction by high-resolution cardiac MRI. Radioinduced toxicity results (pericarditis, myocardial infarction and fatigue) will be classified according to the Common Terminology Criteria for Adverse Events (CTCAE) version 5.0.

All patients will undergo more comprehensive clinical, laboratory and imaging evaluation at 2 time points: up to 2 weeks before and 12 weeks after RT. At each moment, a clinical evaluation will be carried out, blood tests will be checked (blood count and serum levels of urea, creatinine, sodium, potassium, calcium, albumin, magnesium, troponin, creatine kinase MB, C-reactive protein and type B natriuretic peptide) and echocardiography will be performed. Cardiac MRI will be performed just 4 weeks after RT.

Although the risk of late toxicity from RT is low due to the dose administered and high short-term mortality associated with HF itself, all patients will be followed by the research group after the period of additional clinical-laboratory evaluations scheduled in the first 12 weeks after RT. After 12 weeks, all patients will be followed by the research group for clinical-laboratory evaluation every 6 months. Considering the median survival reported in this group of patients, approximately 2 years, the estimated total duration of the study is 5 years.

ELIGIBILITY:
Inclusion Criteria

* Age >18 years;
* Clinical and laboratory diagnosis of chronic systolic HF grades II or III of the New York Heart Association with ejection fraction <40%;
* Refractoriness to standard clinical treatment; defined as the persistence of HF signs and symptoms despite optimized drug therapy.
* Patient consent to participate in the study.
* Agreement to adopt contraceptive practices/methods until the end of the intervention for women of childbearing age.

Exclusion Criteria

* Patients who have undergone any type of previous radiotherapy in the thoracic region;
* Patients who have undergone heart transplants;
* Contraindications for magnetic resonance imaging (MRI), such as the use of metal implants or prostheses.
* Pregnant patients.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2025-07-14 (Estimated); Primary Completion 2025-12-20 (Estimated); Study Completion 2030-09-30 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline in the Left Ventricular Ejection Fraction | 4 weeks after radiotherapy
  Impact of RT on left ventricular ejection fraction by high-resolution cardiac MRI
Treatment-related Adverse Effects as assessed by CTCAE v5.0 | Evaluation at 2, 4, 12 weeks and every 6 months unti 5 years after radiotherapy
  Pericarditis, myocardial infarction and fatigue) will be classified according to the Common Terminology Criteria for Adverse Events (CTCAE) version 5.0.

CONTACTS AND LOCATIONS:
Locations (1):
- Hcor / Associação Beneficente Síria, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Yes
Study Protocol, Statistical Analysis Plan (SAP), Informed Consent Form (ICF), Clinical Study Report (CSR) and Analytic Code
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Six months after the publicationof the article.
Access Criteria: Detailed planned analysis from actives researchers in the topic.